CLINICAL TRIAL: NCT04187872
Title: Recurrent Brain Metastasis Immune Effects and RespOnse to Laser Interstitial ThermotHerapy (LITT) and Pembrolizumab in Combination (TORCH)
Brief Title: LITT and Pembrolizumab in Recurrent Brain Metastasis
Acronym: TORCH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated
Sponsor: University of Florida (Other)
Collaborators: Monteris Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201902411; OCR26353 (Other: UF OnCore)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Melanoma; Non-small Cell Lung Carcinoma (NSCLC); Renal Cell Carcinoma (RCC); Small-cell Lung Cancer; Head and Neck Squamous Cell Cancer; Classical Hodgkin Lymphoma; Primary Mediastinal Large B-Cell Lymphoma; Urothelial Carcinoma; Microsatellite Instability-High Cancer; Gastric Cancer; Esophageal Cancer; Cervical Cancer; Hepatocellular Carcinoma; Merkel Cell Carcinoma; Brain Metastases, Adult
Keywords: Recurrent brain metastases
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Carcinoma, Transitional Cell; Stomach Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Merkel Cell; Brain Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with Recurrent Brain Metastes (Experimental): Adult patients with a primary cancer approved by the FDA for treatment with an immune-checkpoint inhibitor who have recurrent brain metastasis that have failed SRS treatment will receive LITT per standard of care in combination with Pembrolizumab 200mg IV every 3 weeks (+/-3 days) up to 2 years.
  Interventions: Combination Product: LITT + Pembrolizumab

INTERVENTIONS:
Combination Product: LITT + Pembrolizumab — Each patient will undergo brain biopsy and laser interstitial thermotherapy (LITT). As soon as possible, no later than two weeks after LITT, pembrolizumab will be administered via infusion and continue q3wks for up to two years.
  Other Names: NeuroBlate System; Keytruda

SUMMARY:
This is an open-label, historically controlled pilot study investigating the immune effect of Laser Interstitial ThermotHerapy (LITT)+ pembrolizumab in adult patients with a primary cancer approved by the FDA for treatment with an immune-checkpoint inhibitor who have recurrent brain metastasis after prior stereotactic radiosurgery (SRS).

DETAILED DESCRIPTION:
Adult patients with a primary cancer approved by the FDA for treatment with an immune-checkpoint inhibitor who have recurrent brain metastasis that have failed stereotactic radiosurgery treatment will be screened. They will sign consent and complete screening procedures. Each patient will be scheduled to undergo biopsy and LITT treatment. Within two weeks of surgery, patients will begin receiving pembrolizumab every three weeks. Pembrolizumab infusions will continue until brain met recurrence per RANO for Brain Mets or up to two years, whichever comes first. Blood samples will be collected for immune monitoring. Tumor tissue will be collected for immune and genomic studies. Approximately 21 patients will be enrolled to accrue 15 evaluable subjects. Patients will be followed for survival data for one year or until death, whichever comes first.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histologic confirmation of primary cancer approved by the FDA for treatment with an immune-checkpoint inhibitor
2. At least one metastatic lesion has had prior SRS. Each patient's scan must be reviewed by a neurosurgeon or radiation oncologist prior to enrollment.
3. KPS ≥ 70.
4. 18 years or older.
5. Adequate bone marrow and organ function as defined below:

   1. ANC ≥ 1,500/mcL
   2. Platelets ≥ 100,000/mcL
   3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L (transfusion is allowed)
   4. Serum creatinine ≤ 1.5 x IULN OR creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
   5. Serum total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for patients with total bilirubin

   i) 1.5 x IULN f) AST (SGOT) and ALT (SGPT) ≤ 3 x IULN
6. Candidate for pembrolizumab treatment.
7. Candidate for LITT treatment:

   1. Metastatic lesions individually measuring 3.5 cm or less
   2. Only lesions that are growing or new will be treated with LITT
   3. Five (5) or less target metastatic lesions that are new or growing
   4. Lesions accessible with a laser probe as determined by the neurosurgeon performing the procedure
   5. Patient able to undergo MRI scans (no incompatible MRI hardware, etc.)
8. A diagnostic contrast-enhanced MRI of the brain must be performed preoperatively, within 30 days prior to study enrollment.
9. Participants of childbearing age must use effective contraception:

   a) Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Refer to Section 9.3 for guidance on highly effective contraceptive methods.

   i) WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

(1) Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or (2) For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.

b) Males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.

10. Ability of the patient to understand and willingness to sign an IRB approved written informed consent document.

11. Steroid dose equivalent to dexamethasone dose of ≤ 6mg daily at the time of enrollment.

EXCLUSION CRITERIA

1. Actively participating in another clinical trial on active study treatment; follow-up or observational status is acceptable if more than 2 weeks since last study treatment.
2. History of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (with the exception of daily dexamethasone ≤ 6 mg).
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection that will no resolve prior to delivery of treatment (LITT), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
4. History of active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. (Note that prior autoimmune diseases at Grade 1 or 2 per CTCAE v. 4.0 - in the last 2 years that were deemed related to prior use of immunotherapy, will be allowed under this protocol, provided that continuation or subsequent resumption of immunotherapy, regardless of whether systemic treatment had been given, did not result in worsening of signs and symptoms of the aforementioned autoimmune diseases).
5. Pneumonitis within the past 3 years (Note that patients with a history of pneumonitis in the past 3 years that was not aggravated by immunotherapy including immune checkpoint inhibitors or that has clinically resolved or improved and has not recurred or progressed clinically with subsequent immunotherapy including immune checkpoint inhibitors are eligible to participate in the study).
6. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test at screening.
7. Females or males of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 24 weeks after the last dose of study drug.
8. Known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected) infection.
9. Known history of active TB (bacillus tuberculosis).
10. Known history of HIV (HIV 1/2 antibodies).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Immune Effect of LITT plus pembrolizumab | From first dose pembro through 30 days after administration of pembro
  Immune profile of peripheral blood mononuclear cells (PBMCs) as measured by RNA sequencing; analysis will be performed through serial blood draws and will compare each analysis to the patient's baseline prior to treatment.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) of LITT plus pembrolizumab | From first dose pembro to 30 days post final pembro dose
  Adverse events will be collected for each patient from the first dose of pembrolizumab until end of the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Rahman, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - McKnight Brain Institute of the University of Florida, Gainesville, Florida
  - University of Florida Health, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No